CLINICAL TRIAL: NCT07397533
Title: The Effect of Pain Neuroscience Education Added to Aerobic Exercise on Pain, Symptom Severity, and Cortisol Levels in Patients With Irritable Bowel Syndrome
Brief Title: Effects of Aerobic Exercise and Pain Neuroscience Education in Irritable Bowel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IstinyeU-FTR-AD-01
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Aerobic Exercise; Abdominal Pain; Cortisol
MeSH Terms: conditions — Irritable Bowel Syndrome; Abdominal Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study is designed as a parallel-group interventional trial. Participants are allocated to intervention groups and followed concurrently throughout the study period without crossover between groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise Group (Active Comparator): Participants in this group will receive a supervised moderate-intensity aerobic exercise program designed according to the American College of Sports Medicine (ACSM) guidelines. The program will consist of treadmill-based walking sessions performed twice weekly for six weeks. Exercise intensity will be set at 40-59% of Heart Rate Reserve using the Karvonen method, and session duration will be progressively increased.
  Interventions: Behavioral: Exercise
- Aerobic Exercise plus Pain Neuroscience Education Group (Active Comparator): Participants in this group will receive the same aerobic exercise program as the Aerobic Exercise Group. In addition, structured Pain Neuroscience Education sessions will be delivered over a six-week period. The education will address pain neurophysiology, central sensitization, stress responses, safety cues, and cognitive-behavioral strategies aimed at reducing perceived threat related to pain and enhancing engagement in physical activity.
  Interventions: Behavioral: Exercise; Behavioral: Pain Neuroscience Education
- Control Group (No Intervention): Participants in the control group receive standard care and are provided with an informational brochure containing general information related to the condition. No structured exercise program or educational intervention is delivered during the study period.

INTERVENTIONS:
Behavioral: Exercise — Participants will participate in a supervised aerobic exercise program designed according to the American College of Sports Medicine (ACSM) guidelines. The exercise protocol consists of treadmill walking performed three times per week for a total duration of six weeks.
  Each exercise session includes a 5-minute warm-up, 30 minutes of continuous aerobic exercise, and a 5-minute cool-down period. Exercise intensity is individually prescribed at 40-60% of heart rate reserve using the Karvonen formula. Heart rate is monitored throughout the sessions to ensure adherence to the target intensity range.
  All sessions are supervised by a physiotherapist, and exercise progression is adjusted based on participant tolerance and safety considerations.
  Arms: Aerobic Exercise Group; Aerobic Exercise plus Pain Neuroscience Education Group
Behavioral: Pain Neuroscience Education — Pain Neuroscience Education is a structured educational intervention aimed at improving participants' understanding of the neurophysiological mechanisms underlying pain. The education focuses on central sensitization, pain modulation, and the role of the nervous system in chronic pain conditions.
  Educational sessions are delivered by a physiotherapist using standardized verbal explanations and visual educational materials. The content is designed to reduce maladaptive pain beliefs, promote adaptive pain coping strategies, and enhance pain-related knowledge.
  Sessions are conducted regularly throughout the intervention period and are tailored to the participants' comprehension levels while maintaining standardized core educational content.
  Arms: Aerobic Exercise plus Pain Neuroscience Education Group

SUMMARY:
Irritable Bowel Syndrome (IBS) is a chronic disorder of gut-brain interaction characterized by abdominal pain and changes in bowel habits. The aim of this study is to compare the effects of moderate-intensity aerobic exercise alone and aerobic exercise combined with Pain Neuroscience Education on abdominal pain, IBS symptom severity, quality of life, and salivary cortisol levels in individuals with IBS.

Participants will be randomly allocated into three groups: (1) Aerobic Exercise Group, (2) Aerobic Exercise plus Pain Neuroscience Education Group, and (3) Control Group. The aerobic exercise program will consist of supervised walking sessions performed twice weekly for six weeks. Pain Neuroscience Education will be delivered in short, structured sessions over the same six-week period. Assessments will be conducted at baseline and at the end of the intervention. Primary outcomes include abdominal pain intensity, IBS symptom severity, and salivary cortisol levels. Secondary outcomes include quality of life, stool form, and pain-related psychosocial measures. This study aims to provide evidence for non-pharmacological, biopsychosocial approaches in the management of IBS.

DETAILED DESCRIPTION:
This is a single-center, randomized controlled interventional study designed to investigate the added effects of Pain Neuroscience Education (PNE) to aerobic exercise on abdominal pain, symptom severity, and stress-related biological responses in individuals with Irritable Bowel Syndrome (IBS).

IBS is a multifactorial disorder of gut-brain interaction characterized by visceral hypersensitivity, central sensitization, and dysregulation of stress-response systems, particularly the hypothalamic-pituitary-adrenal (HPA) axis. Given the heterogeneous nature of IBS and the limited long-term effectiveness of pharmacological treatments, there is increasing interest in non-pharmacological, biopsychosocial approaches that target both physiological and cognitive-behavioral mechanisms.

Aerobic exercise has been shown to modulate autonomic nervous system activity, inflammatory processes, and stress regulation, which are relevant to IBS symptom expression. Pain Neuroscience Education is a structured educational intervention aimed at reducing perceived threat associated with pain by improving understanding of pain neurophysiology, addressing central sensitization mechanisms, and modifying maladaptive beliefs and avoidance behaviors. The integration of aerobic exercise with PNE is hypothesized to produce more comprehensive and sustainable clinical benefits than exercise alone by simultaneously targeting peripheral, central, and cognitive components of pain.

Adults aged 18-65 years diagnosed with IBS according to Rome IV criteria will be recruited. Participants will be stratified by IBS subtype and sex before being randomly allocated into three study groups.

The aerobic exercise intervention will consist of supervised walking sessions conducted in accordance with the American College of Sports Medicine (ACSM) guidelines. Exercise intensity will be prescribed using the Karvonen heart rate reserve method, targeting 40-59% of heart rate reserve, with progression based on individual tolerance over the six-week intervention period.

Participants allocated to the combined intervention group will receive the same aerobic exercise program along with structured PNE sessions delivered throughout the same six-week period. Educational content will focus on pain neurophysiology, central sensitization, stress responses, safety signaling, pain neuromatrix concepts, and practical coping strategies applicable to daily life.

Participants in the control group will not receive therapeutic exercise or face-to-face education. Instead, they will be provided with standard written information regarding IBS, general pain management principles, and basic recommendations for aerobic physical activity.

This study aims to contribute evidence regarding the role of integrated exercise-based and educational interventions in addressing both clinical symptoms and stress-related mechanisms in the management of IBS.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years
* Diagnosis of Irritable Bowel Syndrome according to Rome IV criteria
* Presence of abdominal pain for at least the past 3 months
* Ability to understand and follow study instructions
* Willingness to participate in the exercise and education sessions
* Provision of written informed consent

Exclusion Criteria:

* Presence of organic gastrointestinal diseases (e.g., inflammatory bowel disease, celiac disease)
* History of gastrointestinal surgery affecting bowel function
* Severe cardiovascular, neurological, or musculoskeletal conditions contraindicating aerobic exercise
* Current participation in a structured exercise program
* Use of medications that may significantly affect gastrointestinal motility or pain perception
* Pregnancy
* Cognitive impairment as indicated by Mini-Mental State Examination score below the cutoff value
* Any medical condition deemed by the investigators to interfere with safe participation in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Abdominal Pain Intensity (Numeric Pain Rating Scale) | Baseline and at the end of the 6-week intervention period
  Abdominal pain intensity is assessed using the Numeric Pain Rating Scale, where participants rate their average abdominal pain intensity over the previous week on an 11-point scale ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain intensity.
IBS Symptom Severity (Irritable Bowel Syndrome Symptom Severity Score) | Baseline and at the end of the 6-week intervention period
  IBS symptom severity will be assessed using the Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS). This validated questionnaire consists of five items evaluating abdominal pain severity, abdominal pain frequency, abdominal bloating, dissatisfaction with bowel habits, and interference of IBS symptoms with daily life.
  Each item is scored from 0 to 100, resulting in a total score ranging from 0 to 500.
  Higher total scores indicate greater IBS symptom severity.
  Symptom severity is commonly categorized as:
  75-174: Mild IBS
  175-299: Moderate IBS
  ≥300: Severe IBS
Salivary Cortisol Level | Baseline and at the end of the 6-week intervention period
  Salivary cortisol levels are measured as a biomarker of physiological stress response. Saliva samples are collected using standardized procedures and analyzed using enzyme-linked immunosorbent assay methods. Cortisol concentrations are normalized to total protein concentration.

SECONDARY OUTCOMES:
IBS-Related Quality of Life (Irritable Bowel Syndrome Quality of Life Questionnaire) | Baseline and at the end of the 6-week intervention period
  IBS-related quality of life will be assessed using the Irritable Bowel Syndrome Quality of Life Questionnaire (IBS-QOL), a disease-specific instrument measuring the impact of IBS on physical, emotional, and social functioning.
  The questionnaire consists of 34 items, with total raw scores ranging from 34 to 170. Raw scores will be transformed to a 0-100 scale, where higher scores indicate better quality of life.
Stool Form (Bristol Stool Form Scale) | Daily during the 6-week intervention period
  Stool form will be assessed using the Bristol Stool Form Scale (BSFS), a validated visual classification system developed by Heaton et al. The scale categorizes stool consistency into seven distinct types.
  Scores range from 1 to 7, where:
  Types 1-2 indicate hard stools associated with constipation,
  Types 3-4 indicate normal stool form,
  Types 5-7 indicate loose or watery stools associated with diarrhea.
  Participants will record stool frequency and form daily throughout the 6-week intervention period. The scale will be used to evaluate IBS symptoms and IBS subtypes.
Pain Catastrophizing (Pain Catastrophizing Scale) | Baseline and at the end of the 6-week intervention period
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS), which evaluates rumination, magnification, and helplessness related to pain experiences.
  Total scores range from 0 to 52, with higher scores indicating greater levels of pain catastrophizing.
Pain Beliefs (Pain Beliefs Scale) | Baseline and at the end of the 6-week intervention period
  Pain-related beliefs will be assessed using the Pain Beliefs Scale (PBS), which evaluates individuals' beliefs regarding the nature, causes, and consequences of pain. The scale consists of 12 items assessing organic and psychological pain beliefs.
  Items are rated on a 1 to 6 Likert scale. Higher subscale scores indicate stronger pain-related beliefs. No cutoff score is defined for this scale.
Pain Knowledge (Revised Neurophysiology of Pain Questionnaire) | Baseline and at the end of the 6-week intervention period
  Pain-related knowledge will be assessed using the Revised Neurophysiology of Pain Questionnaire (RNPQ). The questionnaire consists of 12 items assessing understanding of pain neurophysiology concepts.
  Each correct response is scored as 1, while incorrect or uncertain responses are scored as 0, resulting in a total score ranging from 0 to 12.
  Higher scores indicate greater knowledge of pain neurophysiology.
Physical Activity Level (International Physical Activity Questionnaire - Short Form) | Baseline and at the end of the 6-week intervention period
  Physical activity level is assessed using the International Physical Activity Questionnaire - Short Form, which evaluates walking, moderate-intensity, and vigorous-intensity physical activity over the previous 7 days. Higher scores indicate higher physical activity levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No